CLINICAL TRIAL: NCT03333902
Title: The Comparison Of Different Nerve Blocks For Postoperative Analgesia In Cesarean Delivery: A Randomized Controlled Trial
Brief Title: The Comparison Of Nerve Blocks In Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Feng Xia (Other)
Responsible Party: Sponsor-Investigator, Feng Xia, Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2016]123
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia, Obstetrical
Keywords: quadratus lumborum block; anesthesia; pain, postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QLB type 2 (Experimental): Ultrasound-guided, Inject at the point posterior to quadratus lumborum muscle, 0.2% ropivacaine 30mL in each side for a total of 60mL.
  Subjects also receive an intravenous patient controlled analgesia (PCA) pump of 0.5 mg/mL morphine for 48 hours.
  Interventions: Procedure: QLB; Procedure: Intravenous patient controlled analgesia (PCA)
- QLB type 3 (Experimental): Ultrasound-guided, Inject at the point between the quadratus lumborum and the psoas major muscle, 0.2% ropivacaine 30mL in each side for a total of 60mL.
  Subjects also receive an intravenous patient controlled analgesia (PCA) pump of 0.5 mg/mL morphine for 48 hours.
  Interventions: Procedure: QLB; Procedure: Intravenous patient controlled analgesia (PCA)
- QLB type 2+3 (Experimental): Ultrasound-guided, conduct both QLB type 2 and 3, 0.2% ropivacaine 15mL in each point of injection, for a total of 60mL.
  Subjects also receive an intravenous patient controlled analgesia (PCA) pump of 0.5 mg/mL morphine for 48 hours.
  Interventions: Procedure: QLB; Procedure: Intravenous patient controlled analgesia (PCA)
- epidural anesthesia group (EA) (Active Comparator): Epidural catheter placement was conducted when finishing spinal anesthesia. After surgery, 30 mL saline (placebo) was Injected at the point posterior to the quadratus lumborum in each side for a total of 60mL. We used a single bolus of 0.15% ropivacaine + 2 mg morphine (diluted in 6 ml saline) via epidural cathether.
  Subjects also receive an intravenous patient controlled analgesia (PCA) pump of 0.5 mg/mL morphine for 48 hours.
  Interventions: Procedure: QLB; Procedure: Intravenous patient controlled analgesia (PCA)

INTERVENTIONS:
Procedure: QLB — QLB, quadratus lumborum block.
Procedure: Intravenous patient controlled analgesia (PCA) — Intravenous patient controlled analgesia (PCA) pump was used to supply additional analgesia and removed 48 h post-operationally.

SUMMARY:
The purpose of this study is to investigate the effect of different kinds of popular peripheral nerve blocks for postoperative analgesia after cesarean delivery is completed, compared with traditional epidual analgesia.

DETAILED DESCRIPTION:
Visual Analogue Scale (VAS) and morphine consumption was adopted to evaluate the pain relief.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II
* weight from 50 to 70 kilogrammes
* a normal singleton pregnancy
* ≥37 weeks gestation

Exclusion Criteria:

* congenital coagulopathy
* anatomic abnormalities
* localized skin infection
* allergy to any of the drugs used

Ages: 24 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Subjects undergo cesarean delivery
Enrollment: 102 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
the change trend of Visual Analogue Scale (VAS) at rest and movement | 0-48 hours postoperatively
  The purpose is to view the change of the level of pain assessed by subjects at adjacent time points. We would set 0, 4, 6, 12, 24, 48 hours postoperatively as observational time points.

SECONDARY OUTCOMES:
total morphine consumption | 0-48 hours postoperatively
  total morphine consumption
complications | 0-48 hours postoperatively
  nausea, vomiting, retention of urine, lower limb weakness, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500